CLINICAL TRIAL: NCT06944613
Title: Study of the Usability of an Augmented Reality Exercise for the Cognitive-motor Rehabilitation of Cerebral Palsy (CP) or Acquired Brain Injury (ABI)
Brief Title: Augmented Reality Training for Cerebral Palsy
Acronym: TERAPACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Esquirol (Other)
Responsible Party: Principal Investigator, Julia HAMONET-TORNY, Doctor, Centre Hospitalier Esquirol
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-A00904-41
Record Dates: First submitted 2024-10-23; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Palsy Infantile; Acquired Brain Injury
Keywords: Cognitive rehabilitation; Augmented reality-based programme; Double tasks; Users experiences
MeSH Terms: conditions — Cerebral Palsy; Brain Injuries

STUDY DESIGN:
Intervention Model Description: Cross-sectional pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- exergames (Other): There are two exergames: corsi and zoo games
  Interventions: Device: Augmented reality-based programme/Microsoft Hololens version 2

INTERVENTIONS:
Device: Augmented reality-based programme/Microsoft Hololens version 2 — Participants play two exergames, the aim of this process is to engage cognitive double tasks

SUMMARY:
Rehabilitation programmes for children and adolescents with CP or ABI are not easily accessible, which hinders the development of their physical and cognitive abilities. The Covid-19 pandemic has highlighted the need for specific care for these children and their families. As part of the rehabilitation of these children, it is necessary to offer cognitive-motor or spatial navigation rehabilitation programmes incorporating different sensory stimuli (visual, auditory). In this context, new technologies appear to be a relevant solution for offering fun, personalised rehabilitation with the possibility of remote self-education. Virtual reality is commonly used for paediatric rehabilitation, unlike augmented reality, which is a very recent and promising technology. Before studying the effectiveness of a new augmented reality-based programme, it is essential to assess the usability, user experience, acceptance and potential benefits of this type of device in the cognitive-motor rehabilitation of this population.

The investigators have developed an exergame, using an augmented reality (AR) headset, which will eventually offer a new form of rehabilitation, both fun and interactive, for children and teenagers with CP or ABIs.

Principal Objective:

Assessing the usability of an AR exercise game for children with CP or ABI.

Secondary Objectives:

Evaluating the user experience (attractiveness, emotions) of an AR exergame for children with CP or ABI Evaluating the acceptance of an AR exergame before and after its use in children with CP or ABI To assess the intrinsic motivation associated with AR exercise for CP and ABI children.

To assess the fatigue (mental and physical) associated with exercise in RA in children with CP or ABI.

DETAILED DESCRIPTION:
The study is divided into 3 stages:

* V0 → Pre-inclusion visit carried out during a follow-up consultation (routine care): carried out by the investigator during which a clinical examination to check the inclusion and non-inclusion criteria will be performed. The child and his/her legal guardians are informed of the study (24-hour cooling-off period), and are given a written consent form.
* V1 → Inclusion visit + session 1: Collection of signed consent form and opening of data collection file

The session lasts approximately 2h15 (including breaks) and includes :

i. A pre-session evaluation with : Clinical tests (walking parameters with the helmet (walking speed, step length) + Eyetracking), an acceptance questionnaire before using the device, and a pre-session fatigability scale.

ii. The main body of the session is made up of a phase in which the children familiarise themselves with one of the mini games + a phase of use.

iii. A post-session evaluation with : A questionnaire on usability, user experience, acceptance after using the device, motivation and fatigue after the session.

- V2 → Session 2 (second mini-game): The session lasts approximately 2 hours (including breaks) and includes: i. A pre-session evaluation with : A pre-use acceptance questionnaire and a pre-session fatigue scale ii. The main body of the session is made up of a phase in which the children familiarise themselves with the second mini-game + a phase of use.

iii. A post-session evaluation with : A questionnaire on usability, user experience, acceptance after using the device, motivation and fatigue after the session.

The order of the mini-games is randomised between participants

ELIGIBILITY:
Inclusion Criteria:

* Children with CP or ABI, aged between 10 and 16.
* Children with sufficient listening comprehension skills
* Membership of the French social security system
* Children who have given their consent
* Obligation to obtain written informed consent from legal representatives

Exclusion Criteria:

* Children with a Gross Motor Function Classification System (GMFCS) motor score of over 3
* Children with contraindications to the use of new technologies (e.g. photosensitive epilepsy)
* Children with atypical or uncorrected visual and/or hearing impairment
* Children with unstable medical conditions
* Simultaneous participation in another research protocol that could have an influence on the evaluation of the PLAR system
* Refusal by the child or the family

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
System Usability Scale | Immediately after the intervention
  The children will score 10 statements using a 5-point Likert scale with anchor points at either end ("Strongly disagree" or "Strongly agree"). The scale employs a numerical rating system, with scores ranging from 0 to 100. A score of 85 or above is typically regarded as 'excellent', 75 or above as 'good', and 50 to 75 as 'fair' or 'correct'. A score below 50 indicates a low level of user satisfaction

SECONDARY OUTCOMES:
Semantic user experience | Immediately after the intervention
  This criteria is evaluated with "AttrakDiff" questionnaire. The children will score the 28 items of the questionnaire are in the form of semantic diﬀerentiators (pair of contrasting words) in 7 points (from -3 to 3). The score for each dimension is then analysed. Scores close to the mean (area between -1 and 1) are standard. Scores between 1 and 3 are considered as positive points and between -1 and -3 as negative points of the system.
Emotionnal user experience | Immediately after the intervention
  The user experience of the device will also be assessed using the emotions dimension of the "meCUE" UX scale. Children will rate 8 statements using a 7-point Likert scale with anchor points at either end ("Strongly disagree" or "Strongly agree").
Acceptance | Before and Immediately after the intervention
  Acceptance of the AR device before and after use will be assessed using four dimensions of the Technology Acceptance Model (TAM): perceived usefulness, perceived ease of use, perceived pleasure and behavioural intention to use. Acceptance before use is measured following a short presentation of the device and its purpose (video). The children rated 3 statements per dimension (12 in total) using a 7-point Likert scale with anchor points at either end ("Strongly disagree" or "Strongly agree"). The score for each dimension was then analysed separately.
Motivation | Immediately after the intervention
  Motivation for the session will be measured by the modified "Intrinsic Motivation Inventory" questionnaire. Of the 7 dimensions of this questionnaire, we have chosen 4 (23 items in total) that are of interest to our subject: Interest/Pleasure, Perceived Competence, Effort/Importance, Pressure/Tension. For each item in the 4 dimensions, the children were asked to indicate their agreement using a 7-point Likert scale with anchor points at either end ("Strongly disagree" or "Strongly agree"). The score for each dimension is then analysed separately.
Fatigue | Pre-intervention
  Fatigue (physical and mental) will be measured using the RPE-C "Rating scale of Perceived Exertion for Children", before and after the session. The ratings range from 6 (no fatigue) to 20 (extreme fatigue), accompanied by images of Gaston Lagaffe, representative of the state of fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Julia HAMONEt-TORNY, MD, Principal Investigator — Centre Hospitalier Esquirol
Locations (1):
- Julia HAMONET-TORNY, Limoges, France

IPD SHARING:
Plan to Share IPD: No